CLINICAL TRIAL: NCT05118412
Title: Personal Protein Digestion Variability
Acronym: DiVa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NL 77937.041.21
Record Dates: First submitted 2021-10-29; First posted 2021-11-12 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Digestive System
Keywords: Plant protein; Digestibility; Protein digestion kinetics; Personalized digestibility; Lucerne

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lucerne protein concentrate (Experimental): Lucerne protein concentrate powder presented in the form of a shake.
  Interventions: Other: Lucerne protein concentrate shake
- Whey protein concentrate (Experimental): Whey protein concentrate powder presented in the form of a shake.
  Interventions: Other: Whey protein concentrate shake

INTERVENTIONS:
Other: Lucerne protein concentrate shake — At three out of five test days: Lucerne protein concentrate powder will be mixed with water to obtain a shake, representing a 20g protein load.
  Other Names: Alfalfa protein concentrate shake
  Arms: Lucerne protein concentrate
Other: Whey protein concentrate shake — At two out of five test days: Whey protein concentrate powder will be mixed with water to obtain a shake, representing a 20g protein load.
  Arms: Whey protein concentrate

SUMMARY:
This study aims to quantify the variation in postprandial AA profiles between (and within) individuals after consumption of a poorly digestible plant protein source (Lucerne) and to compare the variation in postprandial AA profiles between a poorly digestible plant protein source and an easy digestible protein source (whey).

The study has a randomised, cross-over, controlled design. Two different treatments, all representing a 20g protein load, will be evaluated on five occasions with a washout period of minimum one week between the test days. On test days, research subjects will receive two different protein sources, in the form of a protein drink, in randomised order; on three test days they will receive a poor-digestible protein source, on two test days an easily digestible protein source. Blood will be collected via a catheter before and up-to four hours after protein consumption. Wellbeing, health complaints or other adverse effects will be collected via short questionnaires during each test day. After each test day gastrointestinal complaints will be collected via an online questionnaire.

DETAILED DESCRIPTION:
There is currently no information on personal protein digestion variability. We recently performed a human intervention study on protein digestibility and absorption and observed that postprandial plasma amino acid (AA) profiles from an easy digestible animal protein were highly comparable among individuals. However, the same profiles from a less digestible plant-protein source (e.g. water lentil) showed a large variability among individuals. But in order to really speak of personalized digestibility, we must be able to demonstrate that the absorption rate of an individual is reproducible. Demonstrating personal differences in AA uptake kinetics will affect the way we value (new) protein sources. Determining and quantifying individual differences in digestion and absorption will allow us to better predict nutritional value of products and diets.

The primary objective is to quantify the variation in postprandial AA profiles between (and within) individuals after consumption of a poorly digestible plant protein source (Lucerne). Secondary objective is to compare the variation in postprandial AA profiles between a poorly digestible plant protein source and an easy digestible protein source (whey).

The study has a randomised, cross-over, controlled design. Two different treatments, all representing a 20g protein load, will be evaluated on five occasions with a washout period of minimum one week between the test days. On test days, research subjects will receive two different protein sources, in the form of a protein drink, in randomised order; on three test days they will receive a poor-digestible protein source, on two test days an easily digestible protein source. Blood will be collected via a catheter before and up-to four hours after protein consumption. Wellbeing, health complaints or other adverse effects will be collected via short questionnaires during each test day. After each test day gastrointestinal complaints will be collected via an online questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women;
* Age between 18 and 40 years;
* Body mass index (BMI) between 18.5 and 30 kg/m2 ;
* Having veins suitable for blood sampling via a catheter (judged by study nurse/ medical doctor).

Exclusion Criteria:

* Any metabolic, gastrointestinal, inflammatory or chronic disease (such as diabetes, anaemia, hepatitis, cardiovascular disease),or having a condition or disease that may lead to an impaired immune system;
* History of gastrointestinal surgery or having (serious) gastrointestinal complaints;
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery;
* Kidney dysfunction (self-reported);
* Any use of medication that may suppress the immune system, this will be judged by the medical supervisor;
* Use of medication that may influence the study results, such as gastric acid inhibitors, laxatives, stomach protectors and drugs that can affect intestinal motility, this will be judged by the medical supervisor;
* Anaemia (Hb values <7.5 mmol/L for women and <8.5 mmol/L for men);
* Reported slimming, medically prescribed or other extreme diets;
* Use of protein supplements;
* Not willing to give up blood donation during the study;
* Current smokers;
* Alcohol intake ≥4 glasses of alcoholic beverages per day;
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported);
* Abuse of hard drugs;
* Not having a general practitioner;
* Participation in another clinical trial at the same time;
* Being an employee of the department Food, Health & Consumer Research of Wageningen Food & Biobased Research or the department of Nutrition and Health of Wageningen University.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Personal variability in 19 amino acid uptake kinetics | Baseline
  Plasma 19 free amino acid levels in venous blood samples under fasting conditions.
Personal variability in 19 amino acid uptake kinetics | 15 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.
Personal variability in 19 amino acid uptake kinetics | 30 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.
Personal variability in 19 amino acid uptake kinetics | 45 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.
Personal variability in 19 amino acid uptake kinetics | 60 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.
Personal variability in 19 amino acid uptake kinetics | 90 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.
Personal variability in 19 amino acid uptake kinetics | 120 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.
Personal variability in 19 amino acid uptake kinetics | 150 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.
Personal variability in 19 amino acid uptake kinetics | 180 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.
Personal variability in 19 amino acid uptake kinetics | 240 minutes post ingestion
  Plasma 19 free amino acid levels in venous blood samples after protein load intake.

SECONDARY OUTCOMES:
Self-reported gastro-intestinal complaints | Before dinner, at the end of each study day
  In order to assess gastro-intestinal complaints, self-reported gastro-intestinal complaints via a online-questionnaire are collected until two days after each test day.
Self-reported gastro-intestinal complaints | Before dinner, first day after each study day.
  In order to assess gastro-intestinal complaints, self-reported gastro-intestinal complaints via a online-questionnaire are collected until two days after each test day.
Self-reported gastro-intestinal complaints | Before dinner, second day after each study day.
  In order to assess gastro-intestinal complaints, self-reported gastro-intestinal complaints via a online-questionnaire are collected until two days after each test day.

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No